CLINICAL TRIAL: NCT04918173
Title: A Multicenter, Prospective, Open-label, Uncontrolled Phase 3 Study to Assess the Efficacy, Safety and Pharmacokinetics of Atenativ in Patients With Congenital Antithrombin Deficiency Undergoing Surgery or Delivery
Brief Title: Efficacy of Atenativ in Patients With Congenital Antithrombin Deficiency Undergoing Surgery or Delivery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN-106
Record Dates: First submitted 2021-05-18; First posted 2021-06-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Congenital Antithrombin Deficiency
MeSH Terms: interventions — Antithrombin III

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atenativ treatment (Experimental): During the PK phase, patients will receive a 60 IU/kg Atenativ as a single intravenous infusion for PK analysis.
  During the treatment phase, patients will receive a single intravenous loading dose followed by maintenance doses administered every 24 hours for approximately 2-7 days for surgical patients and approximately 5 days for parturients
  Interventions: Drug: Atenativ

INTERVENTIONS:
Drug: Atenativ — Antithrombin concentrate

SUMMARY:
The goal of this study is to assess the incidence of the composite of thrombotic events (TEs) and thromboembolic events (TEEs) in patients with congenital antithrombin deficiency under when they receive Atenativ for surgical procedures or parturition.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients ≥18 and ≤80 years of age. Solely in the US, 4 male or female patients between ≥12 and <17 years of age will be enrolled into the PK phase, and subsequently in the treatment phase, if applicable
2. Documented congenital antithrombin deficiency, defined by plasma activity level of antithrombin ≤60% from medical history
3. Personal or family history of TEs or TEEs (except for PK patients)
4. For the Treatment Phase: either a) non-pregnant surgical patients scheduled for elective surgical procedure(s) known to be associated with a high risk for occurrence of TEs or TEEs, or b) pregnant patients of at least 27 weeks gestational age who are scheduled for caesarean section or delivery
5. For female patients of childbearing potential entering the PK Phase who are not known to be pregnant, and for female surgical patients of childbearing potential entering the Treatment Phase for any procedure other than caesarean section or delivery, a negative urine pregnancy test at screening and at baseline
6. Patient has provided informed consent

Exclusion Criteria:

1. Requires emergency surgery or emergency caesarean section
2. Has undergone surgery within the last 6 weeks
3. History or suspicion of another hereditary thrombophilic disorder other than antithrombin deficiency (e.g., activated protein C [APC] resistance/Factor V Leiden, Protein S or C deficiency, prothrombin gene mutation [G20210A], or acquired [lupus anticoagulant] thrombophilic disorder)
4. Malignancies, renal failure (patients on renal replacement therapy), or severe liver disease (aspartate aminotransferase [ASAT] >5 times the upper limit of normal)
5. Body mass index >40 kg/m2 (for non-pregnant patients, only)
6. Known hypersensitivity or allergic reaction to antithrombin or any of the excipients in Atenativ
7. History of anaphylactic reaction(s) to blood or blood components
8. Refusal to receive transfusion of blood-derived products
9. Administration of any antithrombin concentrate or antithrombin-containing blood product within 14 days of either of the two phases of the study
10. Prior diagnosis of heparin-induced thrombocytopenia
11. TE or TEE within the last 6 months
12. Female patients who are nursing at the time of screening*
13. Have participated in another investigational study within the last 30 days
14. Persons dependent on the sponsor, the investigator or the centre of investigation
15. Persons placed in an institution by administrative or judicial order

    * criterion does not include female patients who plan to breastfeed after giving birth

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Thrombotic event incidence | Up to day 30 post treatment initiation
  The primary objective of this study is to assess the incidence of the composite of TEs and TEEs in patients with congenital antithrombin deficiency under cover of Atenativ for surgical procedures or parturition

SECONDARY OUTCOMES:
Single dose Pharmacokinetics of Atenativ: Area under the curve (AUCnorm(0-∞)) | Up to day 14 post PK infusion
  Assess the area under the curve (AUCnorm(0-∞)) of Atenativ in patients with congenital antithrombin deficiency
Single dose Pharmacokinetics of Atenativ: Maximum plasma concentration (Cmax) | Before first infusion, 20 minutes, 1 hour, 3 hours, 8 hrs, 1 day, 2 days, 3, days, 4 days, 5 days, 6 days, 7 days, 8 days, 10 days, 12 days and 14 days post-infusion
  Assess the maximum plasma concentration (Cmax) after a single dose of Atenativ in patients with congenital antithrombin deficiency
Single dose Pharmacokinetics of Atenativ: Half-life (t1/2) | Before first infusion, 20 minutes, 1 hour, 3 hours, 8 hrs, 1 day, 2 days, 3, days, 4 days, 5 days, 6 days, 7 days, 8 days, 10 days, 12 days and 14 days post-infusion
  Assess the half-life (t1/2) after a single dose of Atenativ in patients with congenital antithrombin deficiency
Single dose Pharmacokinetics of Atenativ: Mean residence time (MRT) | Before first infusion, 20 minutes, 1 hour, 3 hours, 8 hrs, 1 day, 2 days, 3, days, 4 days, 5 days, 6 days, 7 days, 8 days, 10 days, 12 days and 14 days post-infusion
  Assess the mean residence time (MRT) after a single dose of Atenativ in patients with congenital antithrombin deficiency
Single dose Pharmacokinetics of Atenativ: Clearance (CL) | Before first infusion, 20 minutes, 1 hour, 3 hours, 8 hrs, 1 day, 2 days, 3, days, 4 days, 5 days, 6 days, 7 days, 8 days, 10 days, 12 days and 14 days post-infusion
  Assess the clearance (CL) after a single dose of Atenativ in patients with congenital antithrombin deficiency
Single dose Pharmacokinetics of Atenativ: Incremental in vivo recovery (IVR) | Before first infusion, 20 minutes, 1 hour, 3 hours, 8 hrs, 1 day, 2 days, 3, days, 4 days, 5 days, 6 days, 7 days, 8 days, 10 days, 12 days and 14 days post-infusion
  Assess the Incremental in vivo recovery after a single dose of Atenativ in patients with congenital antithrombin deficiency
Single dose Pharmacokinetics of Atenativ: Volume of distribution at steady state (Vss) | Before first infusion, 20 minutes, 1 hour, 3 hours, 8 hrs, 1 day, 2 days, 3, days, 4 days, 5 days, 6 days, 7 days, 8 days, 10 days, 12 days and 14 days post-infusion
  Assess the volume of distribution at steady state (Vss) after a single dose of Atenativ in patients with congenital antithrombin deficiency
Single dose Pharmacokinetics of Atenativ: Maximum Plasma Concentration (Tmax) | Before first infusion, 20 minutes, 1 hour, 3 hours, 8 hrs, 1 day, 2 days, 3, days, 4 days, 5 days, 6 days, 7 days, 8 days, 10 days, 12 days and 14 days post-infusion
  Assess the time to reach Maximum Plasma Concentration (Tmax) after a single dose of Atenativ in patients with congenital antithrombin deficiency
10. Coagulation parameters: Activated partial thromboplastin time [aPTT] | Up to day 7 post treatment initiation
  Assess activated partial thromboplastin time [aPTT] in patients with congenital antithrombin deficiency undergoing surgical procedures or parturition
Coagulation parameters: Prothrombin time [PT] | Up to day 7 post treatment initiation
  Assess prothrombin time [PT] in patients with congenital antithrombin deficiency undergoing surgical procedures or parturition
Coagulation parameters: International normalised ratio [INR] | Up to day 7 post treatment initiation
  Assess international normalised ratio [INR] in patients with congenital antithrombin deficiency undergoing surgical procedures or parturition
Coagulation parameters: Fibrinogen level | Up to day 7 post treatment initiation
  Assess fibrinogen in patients with congenital antithrombin deficiency undergoing surgical procedures or parturition
Safety and tolerability: Number of adverse events (AEs) | Up to day 30 post treatment initiation
  Number of adverse events (AEs) following treatment with Atenativ in patients with congenital antithrombin deficiency

CONTACTS AND LOCATIONS:
Locations (30):
- United States (5):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Weill Cornell Medicine, New York, New York
  - Duke University, Durham, North Carolina
- Yeolyan Hematology and Oncology Centre, Yerevan, Armenia
- Universitätsklinik für Innere Medizin Klinische Abteilung für Hämatologie und Hämostaseologie, Vienna, Austria
- Centre for Thrombosis and Haemaostasis, Nymburk, Czechia
- France (3):
  - Centre de Référence de l'Hémophilie Unité d'Hémostase Clinique Hôpital Cardiologique Louis Pradel, Bron
  - University Hospital of Reims, Reims
  - Centre Hospitalier Universitaire de Rouen (CHU de Rouen) - Centre de Traitement des Maladies Hemorragiques (CRTH) (Centre d'Hemophiles), Rouen
- Aversi Clinic, Tbilisi, Georgia
- Germany (3):
  - Klinik fur Angiologie Hamostaseologie Haus 12 A Gerinnungssprechstunde, Berlin
  - UKB Bonn Institut für Experimentelle Hämatologie und Transfusionsmedizin, Bonn
  - Gerinnungszentrum Rhein-Ruhr, Duisburg
- University of Debrecen, Medical and Health Science Centre, Debrecen, Hungary
- Israel (2):
  - Rabin Medical Centre, Institute of Haematology, Petah Tikva
  - Sheba Medical Centre, Ramat Gan
- Italy (4):
  - Unita Strutturale Complessa di Immunoematologia e Medicina Trasfusionale -Dipartimento Interaziendale di Medicina Trasfusionale ed Ematologia - ASST Papa Giovanni XXIII ematologia Piazza OMS, 1, Bergamo
  - Universita degli Studi di Milano - IRCCS Ospedale Maggiore Policlinico - Centro Emofilia e Trombosi Angelo Bianchi Bonomi, Milan
  - University of Padua Medical School, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Emergency County Hospital Craiova, Craiova, Romania
- Clinical Center of Serbia, Belgrade, Serbia
- Spain (4):
  - Central University Hospital of Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Ourense University Hospital, Ourense
- United Kingdom (2):
  - Royal-free Hospital-Katherine Dormandy Haemophilia and Thrombosis Centre, London
  - St. Thomas Hospital, London

IPD SHARING:
Plan to Share IPD: No